CLINICAL TRIAL: NCT01456676
Title: A Single-arm Dose-finding Phase Ib Multicenter Study of the Oral Smoothened Antagonist LDE225 in Combination With Nilotinib in Chronic or Accelerated Phase of Chronic Myeloid Leukemia Patients Who Have Failed Prior Therapy With Other BCR-ABL Tyrosine-kinase Inhibitors
Brief Title: Nilotinib and LDE225 in the Treatment of Chronic or Accelerated Phase Myeloid Leukemia in Patients Who Developed Resistance to Prior Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107Y2101; 2011-000282-12 (EudraCT Number)
Record Dates: First submitted 2011-10-14; First posted 2011-10-21 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-09

CONDITIONS: Philadelphia Chromosome Positive Chronic Myelogenous Leukemia
Keywords: LDE225; nilotinib; Chronic myeloid leukemia; CML; Philadelphia positive; Ph+; resistant; Resistant Philadelphia chromosome positive chronic myeloid leukemia (Ph+ CML) in chronic phase (CP)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; sonidegib

ARMS (1):
- Nilotinib + LDE225 (Experimental): The planned dose of nilotinib 400 mg b.i.d (twice a day) was selected for the combination as this is the dose approved for the treatment of the patient population that will be included in the present study. The starting dose for LDE225 chosen for the current study is 400 mg once daily(q.d.). The maximum dose of LDE225 that will be tested in combination with nilotinib is 800 mg once dail.y
  Interventions: Drug: Nilotinib + LDE225

INTERVENTIONS:
Drug: Nilotinib + LDE225 — Nilotinib is an aminopyrimidine ATP-competitive inhibitor of the protein tyrosine kinaseactivity of BCR-ABL.

SUMMARY:
The purpose of this study is to determine the feasibility of administering the combination of nilotinib and LDE225 to patients with chronic or accelerated phase of chronic myeloid leukemia and to establish the maximum tolerated dose (MTD) and/or recommended Phase II dose level (RP2D) of LDE225 in combination with nilotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Philadelphia chromosome positive (Ph+) CML in chronic phase (CP) or accelerated phase (AP)with resistance to at least one prior BCR-ABL targeting TKI
2. Documented chronic phase CML
3. Adequate end organ function
4. Female patients of childbearing potential must have a negative serum pregnancy test and must be using highly effective methods of contraception. Male patients with female partners of child-bearing potential must use condoms.

Exclusion Criteria:

1. Impaired cardiac function
2. Severe and/or uncontrolled concurrent disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
3. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
4. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to entering the study
5. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either safely discontinued or switched to a different medication prior to starting study drug.
6. Previously documented BCR-ABL Y253H, E255K/V, T315I or F359C/V mutation

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence rate and category of dose limiting toxicities (DLTs) during the first two cycles of therapy | 56 days (2 treatment cycles at 28 days each)
  Determination of the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of nilotinib in combination with LDE225

SECONDARY OUTCOMES:
No of participants with Adverse drug reactions and serious adverse drug reactions, changes in hematology and blood chemistry values, assessments of physical examinations, vital signs and electrocardiograms | 336 days (12 treatment cycles)
  Assessment of the safety and tolerability profile of nilotinib in combination with LDE225
Plasma concentration and basic pharmacokinetics (PK) parameters (as Cmax, Tmax, AUC) | 50 days
  Assessment of the PK characteristics of nilotinib administered in combination with LDE225
Major molecular response (MMR) rates at 3, 6 and 12 months | 336 days (12 treatment cycles)
  Determination of the kinetics of major molecular response
Complete molecular response (CMR) rates at 3, 6 and 12 months | 336 days (12 treatment cycles)
  Determination of the kinetics of complete molecular response
Major cytogenic response (MCyR) rates by 3, 6 and 12 months | 336 days (12 treatment cycles)
  Determination of major cytogenetic response rates
Complete cytogenic response (CCyR) rates by 3, 6 and 12 months | 336 days (12 treatment cycles)
  Determination of complete cytogenetic response rates

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Marseille, France
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Roma, RM, Italy
- Spain (2):
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Madrid

REFERENCES:
- See also: Reuslts for CAMN107Y2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13103